CLINICAL TRIAL: NCT06905691
Title: Effects of Eccentric Training in the Rehabilitation of Patients Undergoing Anterior Cruciate Ligament Reconstruction: a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Bruno Manfredini Baroni, PhD, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 77855224.0.0000.5345
Record Dates: First submitted 2024-04-03; First posted 2025-04-01 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Anterior Cruciate Ligament Reconstruction Rehabilitation; Anterior Cruciate Ligament Reconstruction
Keywords: Knee; Physiotherapy; Quadriceps; Anterior cruciate ligament reconstruction; Eccentric Exercise; Eccentric

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Training Group (Active Comparator): Conventional concentric and eccentric phases
  Interventions: Other: Conventional Training
- Eccentric Training Group (Experimental): Focus on the eccentric phase of movement
  Interventions: Other: Eccentric Training

INTERVENTIONS:
Other: Conventional Training — Patients will execute the concentric and eccentric phases unilaterally, maintaining consistent load levels, with each phase lasting 2 seconds.
  Arms: Conventional Training Group
Other: Eccentric Training — The concentric phase will be performed bilaterally in approximately 1 second, followed by the unilateral eccentric phase lasting approximately 3 seconds.
  Arms: Eccentric Training Group

SUMMARY:
This study aims to investigate the effects of eccentric training on the functional rehabilitation of patients undergoing Anterior Cruciate Ligament Reconstruction (ACL-R). Thirty-four participants undergoing ACL-R will be randomly assigned to two groups: the Conventional Training Group (CTG) and the Eccentric Training Group (ETG). Both groups will adhere to the same post-surgical rehabilitation program, commencing in the first week after ACL-R and continuing until the criteria for sports resumption are achieved. The rehabilitation program will be structured into four phases: immediate post-operative, preparatory, general acquisition, and specific acquisition. The key distinction between the groups lies in their exercise regimen: ETG will prioritize the eccentric phase of movement, whereas CTG will engage in conventional exercises, maintaining uniform load across both movement phases. Assessment procedures will be conducted at three intervals for all participants: immediately post-operative, at 12 weeks post-ACL-R surgery (before the initiation of the training protocol), and at 25 weeks post-ACL-R surgery (upon completion of the training protocol). The primary outcome measure will be the maximum isometric strength of knee extensors. Secondary outcomes will encompass functional status, maximum isometric strength of knee flexors, peak dynamic strength during leg press, quadriceps muscle atrophy, performance in jump tests, and psychological readiness.

ELIGIBILITY:
Inclusion Criteria:

- Individuals of both genders, aged between 18 and 40 years, scheduled for ACL reconstruction surgery during the data collection period.

Exclusion Criteria:

* Delay of more than 7 days after surgery to initiate the rehabilitation program proposed by the study;
* Presence of injuries related to the rupture of the ACL that hinder partial weight-bearing in the first week after surgery, either due to medical recommendation or the patient inability/disposition.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Maximal isometric strength of knee extensors | In the 12th and 25th weeks post-surgery
  Assessed by manual isometric dynamometry

SECONDARY OUTCOMES:
Maximum isometric strength of knee flexors | In the 12th and 25th weeks post-surgery
  Assessed by manual isometric dynamometry
Maximum dynamic strength during leg press exercise | In the 12th and 25th weeks post-surgery
  Assessed through the 1 maximum repetition test (1RM)
Muscle atrophy | In the 12th and 25th weeks post-surgery
  The evaluation of muscle atrophy will be performed by measuring the circumference of the thigh (cm)
Self-reported functional impairments | In the 12th and 25th weeks post-surgery.
  Self-reported functional impairments will be assessed using the International Knee Documentation Committee (IKDC)
Performance in jump tests | In the 12th and 25th weeks post-surgery
  Measured through the Single and Triple Hop Tests
Psychological readiness to return to sport | In the 12th and 25th weeks post-surgery.
  Assessed by Return to Sport after Anterior Cruciate Ligament Reconstruction Surgery (RSI-ACL)

CONTACTS AND LOCATIONS:
Locations (1):
- Private Rehabilitation Center, Veranópolis, Rio Grande do Sul, Brazil